CLINICAL TRIAL: NCT06901635
Title: The Effect Of Dıfferent Cognıtıve Tasks On Manual Dexterıty And Dual Task Performance In Gerıatrıc Indıvıduals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Marmara-OĞUZ-POLAT001
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Dual Task Cost
Keywords: hand dexterity; cognitive function; dual task

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy individuals aged 65-74 years (Other): Box and Block test was used to evaluate the manual dexterity of the participants. Cognitive tasks were given as secondary to the Box and Block test to evaluate the participants' Dual Task performance. In our study, 4 different secondary cognitive tasks were used.
  Interventions: Other: Dual Task
- Healthy individuals aged 75-84 years (Other): Box and Block test was used to evaluate the manual dexterity of the participants. Cognitive tasks were given as secondary to the Box and Block test to evaluate the participants' Dual Task performance. In our study, 4 different secondary cognitive tasks were used.
  Interventions: Other: Dual Task

INTERVENTIONS:
Other: Dual Task — In our study, manual dexterity and cognitive task performance during a dual task will be evaluated. Box and Block Test was used to assess dexterity and 4 different cognitive functions were used as cognitive tasks. Previous studies used one or two cognitive tasks when examining the relationship between cognitive task and dexterity performance during a dual task. This study will examine the effect of different cognitive tasks such as attention, memory, executive functions and working memory on the motor task requiring dexterity during a dual task.

SUMMARY:
Aging is a natural, universal and inevitable process seen in all living things. With aging, structural and functional irreversible degenerative changes occur in molecules, cells, tissues, organs and systems in living organisms. These changes, which extend from cells to systems in aging, may cause limitations in the functions necessary for elderly individuals to maintain their daily life activities such as walking, balance, coordination, visual and auditory skills, cognitive skills and dexterity. WHO defines old age as the period between 65-74 years of age as young old age, 75-84 years of age as middle-aged, and 85 years and older as old age (old age). Manual dexterity is the ability to move an object in a desired manner and is necessary to carry out activities of daily living. Decreases in dexterity may occur with aging, which leads to limitation of activities of daily living. Impaired dexterity leads to a progressive deterioration in the performance of activities of daily living that require the use of the hands. Therefore, the ability of older adults to live comfortably and independently is negatively affected. Numerous factors such as loss of grip strength, sensory disabilities, decreased vision, neuro-muscular problems and cognitive decline can lead to impaired dexterity in older adults. It has been shown that there is a further decline in dexterity with increasing age. One of the reasons affecting manual dexterity in the elderly is cognitive functions. Cognitive functions are a set of functions that enable the perception and understanding of all kinds of inputs received from the sensory organs. These functions include alertness, attention, memory, executive functions, planning, abstraction, language skills, time-space orientation and arithmetic. As with all physiological structures, cognitive functions are also impaired with aging. As age advances, impairments in cognitive functions become more noticeable. The term Dual Task (DT) refers to the ability to perform a cognitive and a motor task simultaneously. The addition of a concurrent cognitive task while performing a motor task often leads to impairment in motor task performance, referred to as the dual task effect (DTE) or dual task cost (DTC). Motor control and executive function are key elements of IG ability, and both are negatively affected by the aging process. Many of the activities of daily living of older adults require dual tasks, such as reading while walking or talking while using cutlery. Therefore, the ability to perform IG is essential for older adults to maintain functional independence. In previous studies, it was observed that when a second cognitive task was given while performing a motor task, motor task and cognitive task decreased; however, the effects of different cognitive tasks on manual dexterity motor task and the difference between young elderly (65-74) and middle-aged (75-84) were not examined. The aim of this study is to examine the effects of cognitive tasks that affect different cognitive functions such as attention, memory and executive functions on the dexterous motor task and to evaluate and compare the differences in two different elderly groups (young and middle-aged). Our study is of great importance in terms of evaluating which cognitive functions are affected during a dual task in elderly individuals and how much dexterity is affected by these functions. Since our study is to obtain data from a certain group in a certain period of time, the type of the research was determined as a cross-sectional study. There are dependent and independent variables in the study. The study aims to examine the effect of different cognitive dual tasks added to a motor task requiring manual dexterity on manual dexterity in geriatric individuals in two different age groups. In this context, the independent variables in the study are the type of cognitive task and age. In total, 4 different cognitive tasks were determined. The dependent variable is dexterity performance. The extent to which dexterity will be affected by 4 different cognitive task types and age will be examined.

ELIGIBILITY:
Inclusion Criteria:

* The participant was determined to be between the ages of 65-84, to be able to cooperate, and to have no obstacle to vision and hearing problems.

Exclusion Criteria:

* The participant had any neurological, rheumatologic and noromuscular disease that would affect the dexterity of the participant, the Mini mental test was below 24, the participant had a hand use problem after any hand injury.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Box and Block Test | 30 second
  The Box and Block Test is a quick, simple and inexpensive test that can be used in various populations to measure unilateral gross manual dexterity. The box and block test consists of a wooden box divided into two compartments by a board and 150 wooden blocks of 2.5 cm3. In the box block test, the person is asked to move the maximum number of blocks one by one from one compartment of the box to the other compartment of equal size within 60 seconds. A trial period of 15 seconds is allowed before starting the test. When placing the blocks in the other compartment, the participant's fingertips must cross the vertical plane of the compartment. The box block test has high reliability in the elderly population. It also has high reliability among manual dexterity assessors and has good criterion construct validity

SECONDARY OUTCOMES:
COGNITIVE TASKS(Executive Functions) | 30 second
  Executive Functions (EF)
  Participants are asked to name animals or fruits and vegetables within a certain time limit. This task has been shown to trigger activation in the frontal network and temporal lobe. This task targets executive function and semantic memory. Participants need to say words, which requires access to their mental lexicon, and they need to focus on the task, select words that meet certain constraints and avoid repetition, which involves executive control processes. Within 30 seconds, the names of animals or vegetables spoken are recorded
COGNITIVE TASK (Working Memory ) | 30 second
  The participant is given a number and asked to count backwards from this number.
  The counting backward task is thought to engage numerical processing skills and is associated with activation in bilateral prefrontal cortices, left posterior inferior perietal lobule and left supementary motor area. The backward counting task is considered a type of mental monitoring that requires retaining information in working memory and mental processing. The counting backward task has been widely used in the literature as a working memory paradigm. Within 30 seconds, the correct numbers spoken are recorded
COGNITIVE TASKS (Attention) | 30 second
  A sequence of numbers is read to the participant. The participant is asked to count the number of times the number is said before the test and to say it at the end of the test.
  Attention can be defined as the ability to selectively process specific information by focusing cognitive resources and ignoring other inputs from the environment. Depending on its tasks, attention can be defined as selective, divided, sustained and shifting attention. The ability to sustain attention is critical for everyday tasks that affect safety, social communication and mental health. Sustained attention is defined as the ability to maintain consistent task performance. This task is a task used to measure sustained attention.
COGNITIVE TASKS(Memory) | 30 second
  The participant is told certain words and then asked to repeat the words back to us. the correct words spoken by the participant are recorded
  This task is used to test short-term memory because the participant is asked to repeat the words immediately after being told them. Episodic memory relies on encoding and retrieval processes and is associated with activation of the bilateral prefrontal cortex. Short-term memory is generally defined as the temporary storage of information. If the information in this structure is encoded or repeated, it is transferred to long-term memory.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"This study does not plan to share individual participant data due to ethical and privacy considerations."